CLINICAL TRIAL: NCT00479999
Title: VRC 012: A Phase I Clinical Trial of the Safety and Immunogenicity of an HIV-1 Adenoviral Vector Serotype 35 Vaccine: Dose Escalation as a Single Agent and Prime-Boost Schedules With an HIV-1 Adenoviral Vector Serotype 5 Vaccine in Uninfected Adults
Brief Title: Phase 1 Safety Study of Two Experimental HIV Vaccines
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 070167; 07-I-0167
Record Dates: First submitted 2007-05-26; First posted 2007-05-30 (Estimated); Last update posted 2019-12-16 (Actual); Status verified 2014-05-05

CONDITIONS: AIDS Vaccines; HIV Infections; HIV-1
Keywords: HIV-Negative; Healthy; Immunity; Preventive; Virus; Healthy Volunteer; HV; HIV Preventive Vaccine
MeSH Terms: conditions — HIV Infections; Virus Diseases

INTERVENTIONS:
Drug: VRC-HIVADV027-00-VP
Drug: VRC-HIVADV038-00-VP

SUMMARY:
This study will test whether two experimental HIV vaccines are safe and whether they cause any side effects in healthy adults. It will examine the body s immune response to the vaccines and monitor the social impact, if any, of being in an HIV vaccine study. The experimental vaccines in this study are the VRC-HIVADV027-00-VP (also called the rAd35-EnvA vaccine) and VRC-HIVADV038-00-VP (also called the rAd5-EnvA vaccine). The vaccines are made using an adenovirus (virus that normally causes respiratory infections and colds) that has been modified to contain DNA that codes for HIV proteins. The vaccines cannot cause HIV or adenoviral infections.

Healthy normal volunteers between 18 and 50 years of age may be eligible for this 2-part study. Part 1 includes 15 people. Part 2 includes 20 people.

Part 1 participants receive only the rAd35-EnvA vaccine. The first five people enrolled receive the lowest study dose of the vaccine. If this dose is safe, then the next five people enrolled receive a higher dose. If this dose is safe, then the last 5 people enrolled receive the highest study dose. Subjects in Part I have about five clinic visits over 24 weeks.

Part II of the study starts after all injections in Part 1 are given. Subjects in Part 2 are randomly assigned to one of two vaccination schedules. One group receives the rAd35-EnvA vaccine first, followed 12 weeks later with the rAd5-EnvA vaccine. The other group receives the vaccines in reverse order; that is, first the rAd5-EnvA vaccine, followed 12 weeks later with the rAd35-EnvA vaccine. In this schedule, the first vaccination primes the immune system and then the immune response is boosted 12 weeks later with a different vaccine. Everyone in study Part 2 receives the rAd35-EnvA vaccine at the middle dose tested in Part 1. Subjects in Part 2 have about eight clinic visits over 36 weeks.

All vaccinations are given as injections in the upper arm. At each clinic visit, participants are checked for health changes or problems. They are asked how they are feeling and if they have taken any medications. Urine samples are collected and blood is drawn at some visits. They are tested for HIV several times and asked questions about their sexual behavior and drug use. Throughout the study, participants are counseled on HIV risk reduction. Subjects are asked about any social effects they may have experienced from their participation in this study.

DETAILED DESCRIPTION:
Study Design:

The VRC recombinant adenoviral vector serotype 5 (rAd5) multiclade vaccine has been previously shown to elicit immune responses to HIV-1-specific peptides when administered intramuscularly (IM) alone and in prime-boost schedules with the greatest magnitude and frequency of response to the Envelope A immunogen (EnvA).

Part I of this study is an open label, dose escalation evaluation of an HIV-1 adenoviral vector serotype 35 vaccine (rAd35-EnvA).

Subjects in Group 1 will receive one vaccination of rAd35-EnvA 10(9) PU.

Subjects in Group 2 will receive one vaccination of rAd35-EnvA 10(10) PU.

Subjects in Group 3 will receive one vaccination of rAd35-EnvA 10(11) PU.

Part II (Group 4) of this study is a randomized, double blind evaluation of the rAd35-EnvA vaccine in comparison to and in combination with a rAd5-EnvA vaccine in prime-boost schedules.

The hypotheses are: 1) rAd35-EnvA vaccine will be safe for human administration at dosages up to 10(11) PU as a single agent and both the rAd35-EnvA and rAd5-EnvA vaccines will be safe in prime-boost regimens; 2) both the rAd35-EnvA and rAd5-EnvA vaccines will elicit immune responses to the EnvA immunogen and 3) the heterologous prime-boost regimens will elicit a greater frequency and magnitude of response than after the priming vaccinations alone. The primary objectives relate to evaluation of the safety and tolerability of the rAd35-EnvA and rAd5-EnvA vaccines. Secondary objectives are related to evaluation of the immunogenicity of the vaccines when comparing rAd35-EnvA to rAd5-EnvA when administered as a prime or as a boost vaccination.

Product Description: Both the VRC-HIVADV038-00-VP (rAd5-EnvA) and the VRC-HIVADV027-00-VP (rAd35-EnvA) vaccines are composed of recombinant, replication deficient adenoviral vectors that encode for HIV-1 clade A Env glycoprotein.

Subjects: Thirty-five healthy adult volunteers, 18 to 50 years old; beginning with the Version 2.0 protocol, subjects in Part I must be Ad35 antibody (Ab) seronegative and subjects in Part II must be both Ad5- and Ad35-seronegative.

Study Plan: Part I: Fifteen subjects will receive an open-label 1 mL IM deltoid injection via needle and syringe of the study agent. No more than one subject per day will be enrolled into each dose group. Five days following vaccination of the fifth volunteer in each dose group, there will be an internal safety review including the principal investigator, clinical team and medical officer to determine whether to proceed to next dose level.

Part II: Initiation of enrollment into Part II will be contingent upon completion of enrollment into Group 3 and a safety review of 10(9) and 10(10) PU dosage by the Data and Safety Monitoring Board (DSMB). The safety review will take place when at least 2 weeks of follow-up on the last 10(10) PU injection in Group 2 is available in the safety reports; the DSMB safety review may occur during enrollment of Group 3.

Enrollment into Group 4 will be randomized and double-blinded. The first 10 subjects in Group 4 will be randomized in a 1:1 ratio into heterologous prime-boost vaccination schedules in which both rAd5-EnvA and rAd35-EnvA are administered at the 10(10) PU dosage. The last 10 subjects in Group 4 will be randomized in a 1:1 ratio into heterologous prime-boost vaccination schedules in which the rAd5-EnvA is administered at 10(10) PU and rAd35-EnvA is administered at 10(11) PU. All subjects will receive each study agent administered as 1 mL IM deltoid injections (12 weeks apart) according to the schedule.

Study Duration

The vaccination regimen and clinical follow-up schedule for Part I requires 24 weeks and for Part II requires 52 weeks to complete. Part II subjects will be contacted annually for 4 years after study completion for collection of long-term follow-up information.

ELIGIBILITY:
* INCLUSION CRITERIA:

A participant must meet all of the following criteria:

1. 18 to 50 years old.
2. Available for clinical follow-up through Week 24 of the study for subjects in Part I: available for clinical follow-up through Week 52 for subjects in Part II and committed to 4 years of annual follow-up contact after Week 52 if in Part II of the study.
3. Able to provide proof of identity to the satisfaction of the study clinician completing the enrollment process.
4. Complete an Assessment of Understanding (that includes understanding of Step Study results) prior to enrollment and verbalize understanding of all questions answered incorrectly.
5. Able and willing to complete the informed consent process.
6. Willing to receive HIV test results and willing to abide by NIH guidelines for partner notification of positive HIV results.
7. Willing to donate blood for sample storage to be used for future research.
8. Willing to discuss HIV infection risks, amenable to risk reduction counseling, committed to maintaining behavior consistent with low risk of HIV exposure through the last required protocol clinic visit and assessed by the clinic staff as being at low risk of HIV infection on the basis of behaviors in the 12 months prior to enrollment as follows:

   Sexually abstinent

   OR

   Had two or fewer mutually monogamous relationships with partners believed to be HIV-uninfected and who did not use injection drugs, crack cocaine or methamphetamine

   OR

   Had three or fewer partners believed to be HIV-uninfected and who did not use injection drugs, crack cocaine or methamphetamine and with whom he/she regularly used condoms for vaginal or anal intercourse.
9. In good general health without clinically significant medical history.
10. Physical examination and laboratory results without clinically significant findings within the 56 days prior to enrollment.

    Laboratory Criteria within 56 days prior to enrollment:
11. Hemoglobin greater than or equal to 11.5 g/dL for women; greater than or equal to 13.5 g/dL for men.
12. White blood cells (WBC) equals 3,300-12,000 cells/mm(3).
13. Differential either within institutional normal range or accompanied by site physician approval.
14. Total lymphocyte count greater than or equal to 800 cells/mm(3).
15. Platelets equal to 125,000 550,000/mm(3).
16. Alanine aminotransferase (ALT) less than or equal to 1.25 times the upper limit of normal.
17. Serum creatinine less than or equal to upper limit of normal (i.e., less than or equal to 1.3 mg/dL for females; less than or equal to 1.4 mg/dL for males).
18. Normal urinalysis defined as negative glucose, negative or trace protein, and no clinically significant blood in the urine.
19. Negative FDA-approved HIV blood test.
20. Negative hepatitis B surface antigen (HBsAg).
21. Negative anti-hepatitis C virus (HCV) antibody and negative HCV PCR.

    Laboratory Criteria within 84 days prior to enrollment:
22. Seronegative for Ad35 antibody if enrolled in Part I after the Version 2.0 amendment and seronegative for both Ad5 and Ad35 antibody if in Part II.

    Female-Specific Criteria:
23. Negative beta-human chorionic gonadotropin pregnancy test (urine or serum) on day of enrollment for women presumed to be of reproductive potential.
24. A female participant must meet any of the following criteria:

No reproductive potential because of menopause [one year without menses] or because of a hysterectomy, bilateral oophorectomy, or tubal ligation,

or

Participant agrees to be heterosexually inactive at least 21 days prior to enrollment and through Week 12 of the study for subjects in Part I and through Week 24 of the study for subjects in Part II,

or

Participant agrees to consistently practice contraception at least 21 days prior to enrollment and through Week 12 of the study for subjects in Part I or through Week 24 of the study for subjects in Part II by one of the following methods:

* condoms, male or female, with or without a spermicide
* diaphragm or cervical cap with spermicide
* intrauterine device
* contraceptive pills or patch, Depo-Provera or other FDA-approved contraceptive method
* male partner has previously undergone a vasectomy.

EXCLUSION CRITERIA:

A volunteer will be excluded if one or more of the following conditions apply:

Women:

1. Woman who is breast-feeding or planning to become pregnant during the 12 weeks of study participation for subjects in Part I and 24 weeks of study participation for subjects in Part II.

   Volunteer has received any of the following substances:
2. HIV vaccine in a prior clinical trial.
3. Immunosuppressive medications, cytotoxic medications, inhaled corticosteroids, or long-acting beta-agonists within the past three months. [With the exceptions that use of corticosteroid nasal spray for rhinitis; topical corticosteroids for an acute uncomplicated dermatitis; short-acting beta-agonists in controlled asthmatics; or a short course (10 days or less) of corticosteroids for a non-chronic condition at least 2 weeks prior to enrollment in this study will not exclude study participation.]
4. Blood products within 120 days prior to HIV screening.
5. Immunoglobulin within 60 days prior to HIV screening.
6. Investigational research agents within 30 days prior to initial study vaccine administration.
7. Live attenuated vaccines within 30 days prior to initial study vaccine administration.
8. Medically indicated subunit or killed vaccines, e.g. influenza, pneumococcal, or allergy treatment with antigen injections, within 14 days of study vaccine administration.
9. Current anti-tuberculosis prophylaxis or therapy.

   Volunteer has a history of any of the following clinically significant conditions:
10. Serious adverse reactions to vaccines such as anaphylaxis, urticaria (hives), respiratory difficulty, angioedema, or abdominal pain.
11. Idiopathic urticaria within the past 2 years.
12. Autoimmune disease or immunodeficiency.
13. Asthma that is unstable or required emergent care, urgent care, hospitalization or intubation during the past two years or that requires the use of oral or intravenous corticosteroids.
14. Diabetes mellitus (type I or II), with the exception of gestational diabetes.
15. History of thyroidectomy or thyroid disease that required medication within the past 12 months.
16. A history of hereditary angioedema, acquired angioedema, or idiopathic forms of angioedema.
17. Hypertension that is not well controlled by medication or blood pressure that is more than 145/95 at enrollment.
18. Bleeding disorder diagnosed by a doctor (e.g., factor deficiency, coagulopathy, or platelet disorder requiring special precautions) or significant bruising or bleeding difficulties with IM injections or blood draws.
19. Within 12 months prior to enrollment: newly-acquired syphilis, gonorrhea, non-gonococcal urethritis, herpes simplex virus type 2 (HSV2), chlamydia, pelvic inflammatory disease (PID), trichomonas, mucopurulent cervicitis, epidiymitis, proctitis, lymphogranuloma venereum, chancroid, or hepatitis B.
20. Malignancy that is active or treated malignancy for which there is not reasonable assurance of sustained cure or malignancy that is likely to recur during the period of the study.
21. Seizure disorder other than: 1) febrile seizures under the age of two, 2) seizures secondary to alcohol withdrawal more than 3 years ago, or 3) a singular seizure not requiring treatment within the last 3 years.
22. Asplenia, functional asplenia or any condition resulting in the absence or removal of the spleen.
23. Psychiatric condition that precludes compliance with the protocol; past or present psychoses; past or present bipolar disorder; disorder requiring lithium; or within five years prior to enrollment, history of a suicide plan or attempt.
24. Any medical, psychiatric, social condition, occupational reason or other responsibility that, in the judgment of the investigator, is a contraindication to protocol participation or impairs a volunteer s ability to give informed consent.
25. BMI greater than or equal to 40; OR BMI greater than or equal to 35 AND with one or more of the following:

    * Age greater than 45
    * Systolic blood pressure greater than 140 mm Hg
    * Diastolic blood pressure greater than 90 mm Hg
    * Current smoker or quit smoking within 28 days of enrollment
    * Untreated or poorly controlled hyperlipidemia
26. Within the 12 months prior to enrollment, one or more of the following:

    * excessive daily alcohol use
    * frequent binge drinking
    * chronic marijuana abuse
    * any other illicit drug use

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2007-05-24; Primary Completion 2014-05-05 (Actual); Study Completion 2014-05-05 (Actual)

PRIMARY OUTCOMES:
Safety (local and systemic reactogenicity, lab tests, AEs)

SECONDARY OUTCOMES:
Immunogenicity (cellular and humoral immune function assays)

CONTACTS AND LOCATIONS:
Overall Officials: Barney S Graham, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Barouch DH, Nabel GJ. Adenovirus vector-based vaccines for human immunodeficiency virus type 1. Hum Gene Ther. 2005 Feb;16(2):149-56. doi: 10.1089/hum.2005.16.149. PMID 15761255
- [Background] Casimiro DR, Chen L, Fu TM, Evans RK, Caulfield MJ, Davies ME, Tang A, Chen M, Huang L, Harris V, Freed DC, Wilson KA, Dubey S, Zhu DM, Nawrocki D, Mach H, Troutman R, Isopi L, Williams D, Hurni W, Xu Z, Smith JG, Wang S, Liu X, Guan L, Long R, Trigona W, Heidecker GJ, Perry HC, Persaud N, Toner TJ, Su Q, Liang X, Youil R, Chastain M, Bett AJ, Volkin DB, Emini EA, Shiver JW. Comparative immunogenicity in rhesus monkeys of DNA plasmid, recombinant vaccinia virus, and replication-defective adenovirus vectors expressing a human immunodeficiency virus type 1 gag gene. J Virol. 2003 Jun;77(11):6305-13. doi: 10.1128/jvi.77.11.6305-6313.2003. PMID 12743287
- [Background] Letvin NL, Huang Y, Chakrabarti BK, Xu L, Seaman MS, Beaudry K, Korioth-Schmitz B, Yu F, Rohne D, Martin KL, Miura A, Kong WP, Yang ZY, Gelman RS, Golubeva OG, Montefiori DC, Mascola JR, Nabel GJ. Heterologous envelope immunogens contribute to AIDS vaccine protection in rhesus monkeys. J Virol. 2004 Jul;78(14):7490-7. doi: 10.1128/JVI.78.14.7490-7497.2004. PMID 15220422
- [Derived] Crank MC, Wilson EM, Novik L, Enama ME, Hendel CS, Gu W, Nason MC, Bailer RT, Nabel GJ, McDermott AB, Mascola JR, Koup RA, Ledgerwood JE, Graham BS; VRC012 Study Team. Safety and Immunogenicity of a rAd35-EnvA Prototype HIV-1 Vaccine in Combination with rAd5-EnvA in Healthy Adults (VRC 012). PLoS One. 2016 Nov 15;11(11):e0166393. doi: 10.1371/journal.pone.0166393. eCollection 2016. PMID 27846256